CLINICAL TRIAL: NCT01555866
Title: A Phase 1 Open Label, 2 Part, Parallel Group Study to Investigate the Effect of Renal Impairment on the Pharmacokinetics of Isavuconazole
Brief Title: Study of the Effect of Renal Impairment on the Pharmacokinetics of Isavuconazole.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Basilea Pharmaceutica International Ltd (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 9766-CL-0018
Record Dates: First submitted 2012-03-14; First posted 2012-03-16 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Pharmacokinetics of Isavuconazole; Healthy Volunteers; Renal Impaired
Keywords: isavuconazole; BAL4815; BAL8557; BAL8728
MeSH Terms: interventions — isavuconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Part 1 Subjects with End Stage Renal Disease (ESRD) (Experimental)
  Interventions: Drug: isavuconazole
- Part 1 Healthy Subjects (Experimental)
  Interventions: Drug: isavuconazole
- Part 2 Subjects with Mild Renal Impairment (Experimental)
  Interventions: Drug: isavuconazole
- Part 2 Subjects with Moderate Renal Impairment (Experimental)
  Interventions: Drug: isavuconazole
- Part 2 Subjects with Severe Renal Impairment (Experimental)
  Interventions: Drug: isavuconazole
- Part 2 Subjects with no Renal Impairment (Experimental)
  Interventions: Drug: isavuconazole

INTERVENTIONS:
Drug: isavuconazole — IV
  Other Names: BAL4815, BAL8557

SUMMARY:
This is a 2-part, open-label study, designed to evaluate the effect of renal disease on the pharmacokinetics of BAL4815 (active isavuconazole moiety) relative to the pharmacokinetics in healthy subjects with normal renal function.

DETAILED DESCRIPTION:
In Part 1, eligible subjects will be enrolled into one of 2 groups based on their renal function. All subjects will receive a single 1-hour infusion of isavuconazole and will remain confined for 4 days. Subjects with normal renal function will return to the clinic for several outpatient visits over 15 days after dosing. Subjects with renal disease will complete the same outpatient visits which correspond to scheduled dialysis dates and then be readmitted to the clinic on study Day 15 to receive a second 1-hour infusion of isavuconazole followed by their normal dialysis procedure and then remain confined for 4 days. ECGs, vital signs, blood draws will be obtained throughout the study for safety and to assess the amount of study drug in the body as well as study drug removed in subjects undergoing dialysis.

In Part 2, eligible subjects will be enrolled into one of 4 groups based on their renal function. All subjects will receive a single 1-hour infusion of isavuconazole and remain confined for 4 days. Subjects will return to the clinic for several outpatient visits over 15 days after dosing. ECGs, vital signs, blood draws will be obtained throughout the study for safety and to assess the amount of study drug in the body.

ELIGIBILITY:
Inclusion Criteria:

* Subject must weigh at least 45 kg and have a body mass index of 18-35 kg/m2
* If female, the subject agrees to sexual abstinence, is surgically sterile, postmenopausal or using a medically acceptable double-barrier method to prevent pregnancy and agrees to continue using this method during the study and until 28 days after final study dug administration. Female subjects must not be lactating or pregnant as documented by a negative pregnancy test at Screening and Day -1
* If male, the subject agrees to sexual abstinence, is surgically sterile, or is using a medically acceptable method to prevent pregnancy and agrees to continue using this method during the study and until 90 days after the end of the study
* The subject has good venous access
* Female subject must not donate ova starting at Screening and throughout the study period, and for 28 days after final study drug administration.

Exclusion Criteria:

* The subject has a previous history of any clinically significant gastro-intestinal, neurological, hepatic, pulmonary, metabolic, dermatologic, immunologic, cardiovascular, psychiatric, genitourinary, endocrine, hematological disorder or disease, malignancy excluding non-melanoma skin cancer or any other medical condition that would preclude participation in the study
* The subject has evidence of any cardiac conduction abnormalities
* The subject has a history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmia, torsade de pointes, structural heart disease, or family history of Long QT syndrome
* The subject has a supine systolic blood pressure less than 90 or greater than 160 mmHg, and diastolic blood pressure less than 50 or greater than 90 mmHg, or pulse rate less than 40 or greater than 100 beats per minute, either at Screening and Day -1
* The subject has a history of consuming more than 14 units of alcoholic beverages per week, has a history of alcohol abuse within the past 2 years prior to Screening, or has a positive screen for alcohol at Screening or Day -1. (NOTE: one unit = 12 ounces of beer, 4 ounces of wine or 1 ounce of spirits/hard liquor.)
* The subject has a positive test for alcohol or drugs of abuse at Screening or Day-1, unless it is an expected result due to an approved concomitant medication for subjects with renal impairment
* The subject has used nicotine patches or any tobacco-containing products within 1 month prior to Day-1 or is a smoker, defined as greater than 10 cigarettes per week
* The subject has had treatment with prescription drugs or complementary and alternative medicines within 14 days prior to Screening, or over-the-counter medication within 14 days prior to Screening (with the exception of acetaminophen up to 2 grams/day)
* The subject anticipates an inability to abstain from caffeine or alcohol for 48 hours prior to Day -1 and throughout the duration of the study
* The subject anticipates an inability to abstain from grapefruit, Seville oranges, star fruit, or any products containing these items from 72 hours prior to Day -1 and throughout the duration of the study
* The subject has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection), or fungal (non-cutaneous) infection within 7 days prior to Day -1
* The subject has been vaccinated within the last 30 days prior to Screening
* The subject has a positive test for hepatitis C antibody or hepatitis B surface antigen at Screening or a known history of human immunodeficiency virus
* The subject has a known or suspected hypersensitivity to isavuconazole, the azole class of compounds, or any components of the study drugs
* The subject has received an experimental agent within 30 days or ten half-lives, whichever is longer, prior to Screening
* The subject has had any significant blood loss, donated one or more units (450 mL) of blood or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days prior to Day -1
* The subject has any other condition, which in the opinion of the investigator, precludes the subject's participation in the trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2012-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics variables for BAL4815 (in plasma): AUC72 and Cmax | Day 1, Part 1
  Area under the concentration-time curve from 0 to 72 hours (AUC72) and Maximum concentration (Cmax)
Pharmacokinetics variables for BAL4815 (in plasma): AUCinf, AUClast, and Cmax | Day 1, Part 2
  Area under the concentration-time curve from time 0 extrapolated to infinity (AUCinf), Area under the plasma concentration-time curve from time of dosing to the last quantifiable concentration (AUClast)

SECONDARY OUTCOMES:
Pharmacokinetics variables for BAL4815 (in plasma): AUCinf and AUClast | Day 1, Part 1
Pharmacokinetics variables for BAL4815 (in plasma): tmax, t1/2, Vz, and CLtot , Ae, Ae% , CLR | Day 1, Parts 1 and 2
  Time to attain maximum concentration (tmax), Apparent terminal elimination half-life (t ½), Apparent volume of distribution during terminal phase (Vz), Total clearance (CLtot), Cumulative amount of unchanged drug excreted in urine (Ae), Percent of drug excreted in urine (Ae%), Renal clearance of the drug from plasma (CLR)
Pharmacokinetics unbound (u) variables for BAL4815 (in plasma and in urine): AUC inf,u, AUC72,u, AUClast,u, Cmax,u, Vz,u, CLtot,u, CLR,u | Day 1, Parts 1 and 2
Pharmacokinetics variables for End Stage Renal Disease (ESRD) subjects for BAL4815: AUC72, Cmax, and tmax | Day 15, Part 1
Pharmacokinetics variables for BAL8728 (in plasma and urine): AUCinf, AUClast, AUC72, Cmax, tmax , t1/2, Vz, CLtot, Ae, Ae% , CLR | Day 1, Parts 1 and 2
Pharmacokinetics variables for End Stage Renal Disease (ESRD) subjects for BAL8728: AUC72, Cmax, and tmax | Day 15, Part 1
Safety assessed by recording adverse events, laboratory assessments, vital signs, electrocardiograms (ECGs) | Part 1: Continuous, up to Day 24; Part 2: Continuous, up to Day 15

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development
Locations (3):
- United States (3):
  - DaVita Research, Denver, Colorado
  - Clinical Pharmacology Miami, Miami, Florida
  - DaVita Clinical Research, Minneapolis, Minnesota